CLINICAL TRIAL: NCT06345261
Title: Role of Diphenhydramine in Prevention of Catheter Related Bladder Discomfort
Brief Title: Diphenhydramine in Catheter Related Bladder Discomfort
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amr Samir Wahdan, Assistant Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2024-872
Record Dates: First submitted 2024-03-28; First posted 2024-04-03 (Actual); Last update posted 2024-04-03 (Actual); Status verified 2024-03

CONDITIONS: Catheter Complications
MeSH Terms: interventions — Diphenhydramine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diphenhydramine group (Active Comparator)
  Interventions: Drug: DiphenhydrAMINE 50 Mg/mL Injectable Solution
- control group (Placebo Comparator)
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: DiphenhydrAMINE 50 Mg/mL Injectable Solution — injection of Diphenhydramine 50 Mg/mL
  Arms: Diphenhydramine group
Drug: Saline — injection of saline
  Arms: control group

SUMMARY:
Diphenhydramine has H1-antihistamine action, it also possesses anti-muscarinic properties. Thus, diphenhydramine might be able to reduce the problem of catheter related bladder discomfort by inhibiting smooth muscle spasm of the urinary bladder via its anti-muscarinic action .

ELIGIBILITY:
Inclusion Criteria:

male patients aged more than18-80 years ASA I and II , upper ureteric stone removal under general anesthesia r

Exclusion Criteria:

overactive bladder cognitive impairment a neuropsychological disorder, bladder outflow obstruction urinary tract infection, , neurogenic bladder, operative time > 6 h

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 104 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-05-01 (Estimated)

PRIMARY OUTCOMES:
incidence of catheter related bladder discomfort postoperative | UP TO 6 HOURE
  * none, did not complain of any CRBD even upon asking.
  * mild, revealed only on questioning.
  * moderate, reported without questioning but not accompanied by any behavioral response.
  * severe, stated on their own and followed by behavioral responses such as a strong verbal response, flailing limbs, and even attempting to pull out the urinary catheter

SECONDARY OUTCOMES:
visual analog scale (VAS) | up to 6 hours
  0 (no pain) to 10 (the worst imaginable pain)

CONTACTS AND LOCATIONS:
Overall Officials: Amr s wahdan, MD, Principal Investigator — Cairo university , Cairo, Egypt
Locations (1):
- Cairo university, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
still working